CLINICAL TRIAL: NCT02242877
Title: Observational Study in Everyday Medical Practice of the Effectiveness of Telmisartan for Treatment of Isolated Systolic Hypertension in Comparison With Systolic/Diastolic Hypertension in Patients Aged 55 or Older
Brief Title: TELSYS - TELmisartan Effectiveness in Isolated SYStolic Hypertension Versus Systolic/Diastolic Hypertension Patients Aged 55 or Older
Acronym: TELSYS
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.510
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Hydrochlorothiazide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Isolated systolic hypertension
  Interventions: Drug: Telmisartan; Drug: Telmisartan combined with hydrochlorothiazide
- Systolic and diastolic hypertension
  Interventions: Drug: Telmisartan; Drug: Telmisartan combined with hydrochlorothiazide

INTERVENTIONS:
Drug: Telmisartan
Drug: Telmisartan combined with hydrochlorothiazide

SUMMARY:
The aim of this study is to compare the effect of treatment with telmisartan on patients in whom the systolic BP is approximately 12 weeks after starting treatment under control for the first time between patients with isolated systolic hypertension (ISH) at the beginning to patients with systolic/diastolic hypertension (SDH)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 55, with no upper limit
* Patient who has been treated and followed up for more than 12 months by the same general practitioner (GP)
* Hypertension measured at least once during the past 12 months and not under control at the time of inclusion in the study:

  * isolated systolic hypertension, namely systolic blood pressure ≥ 140 mmHg and diastolic blood pressure < 90 mmHg or
  * systolic/diastolic hypertension, namely systolic blood pressure ≥ 140 mmHg and diastolic blood pressure ≥ 90 mmHg; or
  * systolic blood pressure ≥ 130 and diastolic blood pressure ≥ 80 mmHg, if the patient has diabetes or chronic renal insufficiency
* Treatment with one or more antihypertensives which remains unchanged during the month prior to collecting the data
* Decision by the GP to add telmisartan (either in combination with hydrochlorothiazide (HCTZ) or not) to the antihypertensive treatment; this decision is made by the treating doctor regardless of participation in the study. The prescription is issued in the normal way, in accordance with the conditions set down in the marketing authorisation
* Written informed consent of the patient to collect his/her data

Exclusion Criteria:

* The patient refuses to allow his/her data to be collected
* Change in the antihypertensive treatment during the month prior to collection of the data
* Blood pressure under control
* The recommended target values corresponding to control of diastolic and systolic blood pressure are important because of the diseases associated with hypertension consequently, and in order to prevent the collection process becoming too complicated, data from patients with severe renal insufficiency or with proteinuria of ≥ 1 g/L or more are not collected in the context of this study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 55 years or older with either isolated systolic- or with systolic and diastolic hyptertension
Sampling Method: Non-Probability Sample
Enrollment: 3320 (Actual)
Dates: Start 2006-02; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Normalization of arterial systolic hypertension | Up to 12 weeks after start of treatment

SECONDARY OUTCOMES:
Assessment of systolic blood pressure (SBP) response | Up to 12 weeks after start of treatment
Mean decrease in systolic blood pressure | Up to 12 weeks after start of treatment
Number of patients with adverse events | Up to 12 weeks